CLINICAL TRIAL: NCT05863351
Title: Phase III Randomized Trial of Stereotactic Ablative Radiotherapy (SAbR) for Oligometastatic Advanced Renal Carcinoma (SOAR)
Brief Title: Focused Radiation Versus Systemic Therapy for Kidney Cancer Patients With Limited Metastasis, SOAR Study
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA8211; NCI-2023-02060 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA8211 (Other: ECOG-ACRIN Cancer Research Group); EA8211 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2023-05-08; First posted 2023-05-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Renal Cell Carcinoma; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (usual care) (Active Comparator): Patients receive standard of care systemic therapy on study. Patients undergo CT or MRI throughout the trial.
  Interventions: Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Procedure: Systemic Therapy
- Arm II (SAbR, usual care) (Experimental): Patients undergo repeated SAbR until progression and then receive standard of care systemic therapy on study. Patients undergo CT or MRI throughout the trial.
  Interventions: Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Procedure: Stereotactic Ablative Radiotherapy; Procedure: Systemic Therapy

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Other: Questionnaire Administration — Ancillary studies
Procedure: Stereotactic Ablative Radiotherapy — Undergo SAbR
  Other Names: SABER; SABR/SBRT
  Arms: Arm II (SAbR, usual care)
Procedure: Systemic Therapy — Given standard of care systemic therapy

SUMMARY:
This phase III trial compares the effect of stero-ablative radiotherapy (SAbR) followed by standard of care systemic therapy, to standard of care systemic therapy alone, in patients with kidney cancer that has spread from where it first started (primary site) to a limited (2-5) number of places in the body (metastatic). Study doctors want to find out if this approach is better or worse than the usual approach for metastatic kidney cancer. The usual approach is defined as the care most people get for metastatic kidney cancer which includes systemic therapy such as immunotherapy (given through the veins) and/or small molecular inhibitor (tablets taken by mouth). Radiotherapy uses high energy x-rays to kill cancer cells and shrink tumors. SAbR uses special equipment to position a patient and deliver radiation to tumors with high precision. Giving SAbR prior to systemic therapy may kill more tumor cells than the usual approach, which is systemic therapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare overall survival (OS) between patients receiving SAbR + systemic therapy (SABR+ST) versus systemic therapy (ST) only.

II. To compare average adverse event (AE) score between SAbR+ST arm and ST only arm.

SECONDARY OBJECTIVES:

I. To compare global health status / quality of life (QOL) between patients receiving SAbR+ST versus ST only.

II. To compare progression-free survival (PFS) between the arms.

EXPLORATORY OBJECTIVES:

I. To estimate PFS on first line systemic therapy (PFS-SST) in the SAbR+ST arm and compare with first line systemic therapy PFS of the ST arm.

II. To explore local control from SAbR by looking at the amount of local failures after SAbR in the SAbR+ST arm.

III. To assess the cost-effectiveness between the arms in terms of cost per unit gain in quality-of-life years.

QOL OBJECTIVES:

I. To compare global health status / quality of life (QOL) between patients receiving SabR+ST versus ST only using the National Comprehensive Cancer Network (NCCN) / Functional Assessment of Cancer Therapy Kidney Cancer Symptom Index -19 item (NFKSI-19).

II. To compare quality-adjusted survival between patients randomized to receive SabR+ST vs ST alone using European Quality of Life (EUROQOL) 5-dimension, 5-level (EQ-5D-5L) at 3, 6, 9, 12, 18, and 24 months.

III. To compare global health status / QOL of the NFKSI-19 at all of the 3, 6, 9, 12, 18, and 24 month time points between patients randomized to receive SabR+ST versus ST alone.

IV. To compare scale scores of the NFKSI-19 (disease-related symptoms - physical disease-related symptoms - emotional, treatment side effects, and function & well-being) at 3, 6, 9, 12, 18, 24 months between patients randomized to receive SabR+ST versus ST alone.

V. To compare time to global quality of life deterioration between patients randomized to receive SabR+ST versus ST alone using NFKSI-19.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard of care systemic therapy on study.

ARM II: Patients undergo repeated SAbR until progression and then receive standard of care systemic therapy on study.

Patients in both arms undergo computed tomography (CT) or magnetic resonance imaging (MRI) throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be >= 18 years of age
* Patient must have a pathologically (histologically or cytologically) proven diagnosis of renal cell carcinoma (RCC) prior to randomization
* Patient may have any RCC histology except a histology that has a sarcomatoid component
* Patient must have primary site addressed by local therapy. If the primary RCC is intact, the patient must undergo local treatment to the primary before randomization
* Patient must have favorable or intermediate International Metastatic RCC Database Consortium (IMDC) risk (0-2) at the time of randomization
* Patient must have a total of between 2 and 5 metastatic lesions, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria with imaging obtained within 45 days prior to randomization
* Patient must have a documentation from a radiation oncologist confirming that all sites are amenable to SAbR
* Patient may have received prior therapy in the adjuvant setting as long as potential trial participants have recovered from clinically significant adverse events of their most recent therapy/intervention prior to enrollment
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* All patients of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy

  * A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria:

    * Has achieved menarche at some point
    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible
* Patient must have a Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Patients must have adequate organ and bone marrow function as per the recommended guidelines and the respective Food and Drug Administration [FDA] package insert required for the systemic therapy chosen by the treating oncologist. We recognize that patients may have varying levels of renal and liver function that will impact which systemic therapy is appropriate for the patient. We do not require all patients to have specific baseline laboratory thresholds but do ask the treating oncologist to attest that the patient has adequate organ and bone marrow function to safely receive one of the first line systemic therapies listed in the protocol as a standard of care treatment option
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial. Testing for HIV is not required for entry onto the study
* For patients with history of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. If no previous history, testing for HBV is not required for entry onto the study
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load. If no previous history, testing for HCV is not required for entry onto the study
* In order to participate in the QOL portion of the protocol, the patient must speak one of the languages in which the NFKSI-19 and EQ-5D-5L is available

  * NOTE: Sites cannot translate the associated QOL forms

Exclusion Criteria:

* Patient must not have brain metastases
* Patient must not have metastasis involving the following locations: ultra-central (within 2cm of carina) lung, invading gastrointestinal tract (such as esophagus, stomach, intestines, colon, rectum), skin, and scalp
* Patient must not have received any prior systemic therapy (except for adjuvant setting) for metastatic RCC
* Active autoimmune disease requiring ongoing therapy including systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications daily. Inhaled steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* History of severe allergic, anaphylactic or other hypersensitivity reactions to chimeric or humanized antibodies
* Active tuberculosis (purified protein derivative [PPD] response without active TB is allowed)
* Uncontrolled hypertension (systolic blood pressure [BP] > 190mmHg or diastolic BP > 110mmHg)
* Major surgery within 30 days prior to randomization
* Any serious (requiring hospital stay or long term rehab) non-healing wound, ulcer, or bone fracture within 30 days prior to randomization
* Any arterial thrombotic (ST elevation myocardial infarction [STEMI], non-STEMI [NSTEMI], cerebrovascular accident [CVA], etc.) events within 180 days prior to randomization
* Moderate or severe hepatic impairment (child-Pugh B or C)
* Untreated pulmonary embolism (PE) or deep-vein thrombosis (DVT) is not allowed. Treated PE or DVT is allowed > 30 days from diagnosis and when not resulting in respiratory impairment
* Unstable cardiac arrhythmia within 180 days prior to randomization
* History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, bowel obstruction, or gastric outlet obstruction within 180 days prior to randomization
* History of or active inflammatory bowel disease
* Malabsorption syndrome within 30 days prior to randomization
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used
* Patient must not expect to conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study and for 6 months after the last dose of protocol treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2037-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization to death from any cause, assessed up to 10 years
  The repeated confidence interval method will be utilized. At each scheduled interim analysis, a one-sided 95% repeated confidence interval of hazard ratio (stereotactic ablative radiotherapy [SAbR] + standard therapy [ST] / ST) will be computed, using the partial likelihood estimate, to test non-inferiority in OS for SAbR+ST arm.
Incidence of adverse events (AEs) | From randomization up to 6 months
  All patients who receive treatment, regardless of eligibility, will be evaluated for AE/toxicity. AE score will be calculated in 3-month intervals starting from randomization. To calculate the AE score for a 3-month interval, for each patient, the AE sub-score for each Common Terminology Criteria for Adverse Events (CTCAE) categories (there are 26 AE categories listed in CTCAE version 5) will be aggregated based on the highest grade of AE experienced in each CTCAE category.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From randomization to progression of disease, assessed up to 10 years
  Patients randomized to SAbR will need to first progress on SAbR, then progress on systemic therapy to be counted as an event for progression. Progression on SAbR is when SAbR (sequential SAbR) is unable to control the disease by meeting one of the two criteria: > 6 metastases in total requiring SAbR (no matter how many metastases a patient was randomized with), or one or more progressing lesions not amenable to SAbR (> 5% risk of grade 3 toxicity by American Society for Therapeutic Radiology and Oncology definition). This endpoint will be compared between the two arms using stratified log-rank test, at one-sided 0.025 significance level.

OTHER OUTCOMES:
PFS-start of systemic therapy (SST) | From the start of SST to progression or death, assessed up to 10 years
  Compare the PFS from the start of systemic therapy (instead of from the time of randomization) of Arm A (after PFS-SAbR) with PFS of upfront systemic therapy in Arm B. This endpoint will be descriptive and will only be explored in arm A. Will explore local control that SAbR provides, by looking at local failures after SAbR in SAbR+ST arm only. Local failure is defined as > 30% increase in the longest diameter of SAbR-treated lesion, more than 6 months post SAbR treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Raquibul Hannan, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (108):
- United States (108):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Mission Cancer and Blood - Ankeny, Ankeny, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mission Cancer and Blood - West Des Moines, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Lenox Hill Hospital, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin